CLINICAL TRIAL: NCT01735721
Title: Comparative Study of Algipore and Decalcified Freeze-dried Bone Allograft in Open Maxillary Sinus Elevation Using Piezoelectric Surgery
Brief Title: Comparative Study of Algipore and Decalcified Freeze-dried Bone Allograft in Open Maxillary Sinus Augmentation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Moeintaghavi, Professor of Periodontics, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 86319
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Disorder of Maxillary Sinus; Maxillary Sinus Floor Augmentation
Keywords: Sinus Floor Augmentation; Bone Transplantation; Bone Substitute

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Sinus Lift with DFDBA (Active Comparator): In each patient, one sinus was chosen at random and filled with DFDBA (Tissue Regeneration Corporation, Iran).
  Interventions: Procedure: Open Sinus Lift
- Open Sinus Lift with Algipore (Experimental): The contra lateral sinus was filled with Algipore (Dentsply, USA).
  Interventions: Procedure: Open Sinus Lift

INTERVENTIONS:
Procedure: Open Sinus Lift — A crestal incision was made on the mucosa of the edentulous ridge. The flap was elevated carefully and extended labially to expose the bone. A vertical releasing incision was made in the mesial end of the flap as needed. The mucoperiosteal flap was extended to expose the alveolar ridge and the lateral wall of the maxillary sinus. Then, a window was prepared using the piezoelectric device (Mectron, Italy); the Schneiderian membrane was then elevated conservatively according to the technique described by Vercellotti (2001).
  The sinus membrane was meticulously detached and pushed superiorly to allow for the placement of bone graft material.

SUMMARY:
The aim of this study was the radiographic and clinical comparison of Algipore with decalcified freeze-dried bone allograft (DFDBA) in the open maxillary sinus lift technique using piezoelectric instruments.

DETAILED DESCRIPTION:
Vertical and horizontal bone resorption of the alveolar ridge are common in edentulous jaws. In the distal area of the maxilla, an adequate bone volume is often lacking because of the proximity of the sinus cavities to crestal bone. Sinus floor augmentation is an established way of increasing the height and volume of bone in the posterior region of the maxilla, which increase the stability of dental implants. For this purpose various materials, including auto grafts, allografts, alloplasts, and xenografts have been used.

ELIGIBILITY:
Inclusion Criteria:

* physically healthy patients
* ridge bone height of less than 5 mm

Exclusion Criteria:

* any past medical history of systemic or localized diseases that were contraindications for sinus or implant surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
increase in bone height | 9 months
  Baseline and 9 months radiographs were scanned with an Agfa scanner at 1200 dpi with a 12-bit grayscale and stored in JPEG format. Changes in bone height were calculated in each case. Two reference points, one at the lowest part of the ridge crest and the other at the highest part of sinus floor, were selected in two radiographs (baseline and after 9 months) and their distance was calculated in 0.1mm scale using computer.

SECONDARY OUTCOMES:
Bone Density | 9 months
  Changes in radiographic density after sinus grafting were evaluated using densitometry.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moeintaghavi, DDS., Msc., Study Director — Mashhad University of Medical Sciences
Locations (1):
- Amir Moeintaghavi, Mashhad, Khorasan Razavi, Iran